CLINICAL TRIAL: NCT03743038
Title: A Randomized, Evaluator-Blinded, Bilateral Comparison Study of Two Topicals in the Treatment of Subjects With Acne Vulgaris
Brief Title: A Study Comparing Two Topicals in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FX2018-23
Record Dates: First submitted 2018-11-10; First posted 2018-11-15 (Actual); Results first posted 2021-02-23 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Minocycline; Ethanol; Solutions

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomized (1:1) to treatment with Test Article A to one side of the face versus Test Article B on the contralateral side.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FMX101 vehicle (Experimental): FMX101 hydrophobic oil based vehicle (Test Article A) topically applied daily for six weeks on one side of the face (in a split-face model)
  Interventions: Drug: FMX101 vehicle
- Hydro-alcohol solution base (Experimental): Hydro-alcohol solution based vehicle (Test Article B) topically applied daily for six weeks on the contralateral side of the face (in a split-face model)
  Interventions: Other: Hydro-alcohol solution

INTERVENTIONS:
Drug: FMX101 vehicle — FMX101 vehicle - hydrophobic oil based vehicle (Test Article A)
  Other Names: Test Article A
  Arms: FMX101 vehicle
Other: Hydro-alcohol solution — Hydro-alcohol solution based vehicle (Test Article B)
  Other Names: Test Article B
  Arms: Hydro-alcohol solution base

SUMMARY:
A Randomized, Evaluator-Blinded, Bilateral Comparison Study to Evaluate the Safety and Efficacy of Two Topicals in the Treatment of Subjects With Acne Vulgaris (Study FX2018-23).

DETAILED DESCRIPTION:
A Randomized, Evaluator-Blinded, Bilateral Comparison Study to Evaluate the Safety and Efficacy of Two Topicals in the Treatment of Subjects With Acne Vulgaris. Eligible subjects will be randomized (1:1) to treatment with Test Article A to one side of the face versus Test Article B on the contralateral side.

ELIGIBILITY:
Inclusion Criteria:

* Has facial acne vulgaris with:

  16 inflammatory lesions (papules, pustules) The inflammatory lesion count on the right and left side of the face should be similar IGA score of moderate (3) on both the right and left side of the face

Exclusion Criteria:

* Acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne), or any dermatological condition of the face or facial hair (eg, beard, sideburns, mustache) that could interfere with the clinical evaluations.
* More than two facial nodules/cysts
* Sunburn on the face

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Site #01, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted in one site at United States from November 20, 2018 to February 11, 2019.
Pre-assignment Details: The study consisted of a Screening/Baseline Visit, Visits at Weeks 1, 2, and 4, along with a Week 6/End of Treatment (EOT) Visit, and a Week 7/End of Study (EOS) Visit. All participants underwent inclusion and exclusion criteria assessment and all eligible participants signed the informed consent before undergoing any study related procedures. All assessments at screening were done as per the schedule of assessment.
Units Other Than Participants: Face sides
Groups:
- Overall: Participants were randomized (1:1) and applied FMX101 hydrophobic oil based vehicle (Test Article A) topically on one side of the face and Hydro-alcohol solution based vehicle (Test Article B) on the contralateral side of the face once daily for six weeks.
Period: Overall Study
Arm/Group | Overall
Started (Test Article A and Test Article B) | 12; 24 Face sides
Test Article A | 12; 12 Face sides
Test Article B | 12; 12 Face sides
Completed (Test Article A and Test Article B) | 11; 22 Face sides
Not Completed | 1; 2 Face sides
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population included all randomized participants who met all Inclusion/Exclusion criteria, applied at least one dose of test article, and returned for at least one post-Baseline evaluation visit.
Groups:
- Overall: Participants were randomized (1:1) and applied FMX101 hydrophobic oil based vehicle (Test Article A) topically on one side of the face and Hydro-alcohol solution based vehicle (Test Article B) on the contralateral side of the face once daily for six weeks on one side of the face.
Arm/Group | Overall
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.1 (5.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 0 to 4 Investigator's Global Assessment Score at Week 6
Description: Severity of acne vulgaris was assessed by Investigator Global Assessment (IGA). The IGA score is a static evaluation of the overall severity or "average" degree of severity of a participant's disease by the Blinded Evaluator taking into account all of the participant's facial acne lesions as the participant appears on the day of the evaluation. Overall severity of acne was assessed using a five-point scale where 0=Clear, 1=Almost Clear, 2=Mild, 3=Moderate, and 4=Severe. Low score represented best outcome and higher score value indicated worst outcome.
Time Frame: At Week 6
Population: The mITT population included all randomized participants who met all Inclusion/Exclusion criteria, applied at least one dose of test article, and returned for at least one post-Baseline evaluation visit. Here, overall number of participants analyzed presents only those participants who were analyzed for this particular outcome measure, and number analyzed presents the number of participants that were analyzed at specified week.
Measure: Number; unit: Participants
Units Other Than Participants: Face sides
Groups:
- FMX101 Oil Vehicle (A): Participants applied FMX101 hydrophobic oil based vehicle (Test Article A) topically once daily for six weeks on one side of the face.
- Hydro-alcohol Vehicle (B): Participants applied Hydro-alcohol solution based vehicle (Test Article B) topically once daily for six weeks on the contralateral side of the face.
Arm/Group | FMX101 Oil Vehicle (A) | Hydro-alcohol Vehicle (B)
Number analyzed (Participants) | 10 | 10
Number analyzed (Face sides) | 10 | 10
Participants
  0-Clear | 0 | 0
  1-Almost Clear | 3 | 3
  2-Mild | 5 | 3
  3-Moderate | 3 | 5
  4-Severe | 0 | 0

2. Primary Outcome: Number of Participants Achieving Investigator's Global Assessments Treatment Success at Week 6
Description: Severity of acne vulgaris was assessed by IGA. The IGA score is a static evaluation of the overall severity or "average" degree of severity of a participant's disease by the Blinded Evaluator taking into account all of the participant's facial acne lesions as the participant appears on the day of the evaluation. Overall severity of acne was assessed using a five-point scale where 0=Clear, 1=Almost Clear, 2=Mild, 3=Moderate, and 4=Severe. The IGA treatment "success" was defined as at least a two-point improvement in IGA score relative to Baseline.
Time Frame: At Week 6
Population: The mITT population included all randomized participants who met all Inclusion/Exclusion criteria, applied at least one dose of test article, and returned for at least one post-Baseline evaluation visit. Here, overall number of participants analyzed presents only those participants who were analyzed for this particular outcome measure.
Measure: Number; unit: Participants
Units Other Than Participants: Face sides
Arm/Group | FMX101 Oil Vehicle (A) | Hydro-alcohol Vehicle (B)
Number analyzed (Participants) | 10 | 10
Number analyzed (Face sides) | 10 | 10
Participants | 3 | 3

3. Primary Outcome: Absolute Change From Baseline to Week 6 in Inflammatory Lesion Count
Description: Inflammatory lesion count (ILC) included papules (raised inflammatory lesions with no visible purulent material) and pustules (raised inflammatory lesions with visible purulent material).
Time Frame: Day 1/ Baseline and Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Lesions
Units Other Than Participants: Face sides
Arm/Group | FMX101 Oil Vehicle (A) | Hydro-alcohol Vehicle (B)
Number analyzed (Participants) | 10 | 10
Number analyzed (Face sides) | 10 | 10
Lesions | -7.5 (8.26) | -6.3 (4.20)

4. Primary Outcome: Percentage Change From Baseline to Week 6 in Inflammatory Lesion Count
Description: The ILC included papules (raised inflammatory lesions with no visible purulent material) and pustules (raised inflammatory lesions with visible purulent material).
Time Frame: Day 1/ Baseline and Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Units Other Than Participants: Face sides
Arm/Group | FMX101 Oil Vehicle (A) | Hydro-alcohol Vehicle (B)
Number analyzed (Participants) | 10 | 10
Number analyzed (Face sides) | 10 | 10
Percent Change | -37.7 (42.88) | -39.0 (30.83)

5. Primary Outcome: Absolute Change From Baseline to Week 6 in Non-Inflammatory Lesion Count
Description: The non-inflammatory lesion count (NILC) included open and closed comedones.
Time Frame: Day 1/ Baseline and Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Lesions
Units Other Than Participants: Face sides
Arm/Group | FMX101 Oil Vehicle (A) | Hydro-alcohol Vehicle (B)
Number analyzed (Participants) | 10 | 10
Number analyzed (Face sides) | 10 | 10
Lesions | -7.0 (5.06) | -5.0 (4.36)

6. Primary Outcome: Percentage Change From Baseline to Week 6 in Non-Inflammatory Lesion Count
Description: The NILC included open and closed comedones.
Time Frame: Day 1/ Baseline and Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Units Other Than Participants: Face sides
Arm/Group | FMX101 Oil Vehicle (A) | Hydro-alcohol Vehicle (B)
Number analyzed (Participants) | 10 | 10
Number analyzed (Face sides) | 10 | 10
Percent Change | -33.2 (24.65) | -24.0 (24.15)

7. Primary Outcome: Change in Sebum Percentage Relative to Baseline Versus Weeks 2, 4, 6 and 7
Description: Sebum measurement was conducted on the right and left side of the face. The sebum measurement represented the sebum score of saturation of the film and had a range of 0 to 99, where 99 equated to very oily skin.
Time Frame: Day 1/Baseline and Weeks 2, 4, 6 and 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage (%)
Units Other Than Participants: Face sides
Arm/Group | FMX101 Oil Vehicle (A) | Hydro-alcohol Vehicle (B)
Number analyzed (Participants) | 12 | 12
Number analyzed (Face sides) | 12 | 12
Percentage (%)
  Week 2: number analyzed (Participants) | 11 | 11
  Week 2: number analyzed (Face sides) | 11 | 11
  Week 2 | 1.6 (13.28) | -2.5 (5.89)
  Week 4: number analyzed (Participants) | 9 | 9
  Week 4: number analyzed (Face sides) | 9 | 9
  Week 4 | 6.0 (13.96) | 5.2 (8.14)
  Week 6: number analyzed (Participants) | 10 | 10
  Week 6: number analyzed (Face sides) | 10 | 10
  Week 6 | 3.9 (8.88) | 1.9 (5.63)
  Week 7: number analyzed (Participants) | 11 | 11
  Week 7: number analyzed (Face sides) | 11 | 11
  Week 7 | -1.9 (8.24) | -1.5 (7.57)

8. Primary Outcome: Change in Transepidermal Water Loss Relative to Baseline Versus Weeks 2, 4, 6 and 7
Description: Transepidermal Water Loss (TEWL) was conducted on the right and left side of the face.
Time Frame: Day 1/Baseline and Weeks 2, 4, 6 and 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/m^2 /h
Units Other Than Participants: Face sides
Arm/Group | FMX101 Oil Vehicle (A) | Hydro-alcohol Vehicle (B)
Number analyzed (Participants) | 11 | 11
Number analyzed (Face sides) | 11 | 11
g/m^2 /h
  Week 2: number analyzed (Participants) | 10 | 10
  Week 2: number analyzed (Face sides) | 10 | 10
  Week 2 | 2.8 (7.12) | -0.4 (5.62)
  Week 4: number analyzed (Participants) | 8 | 8
  Week 4: number analyzed (Face sides) | 8 | 8
  Week 4 | 1.3 (6.86) | -1.2 (6.46)
  Week 6: number analyzed (Participants) | 10 | 10
  Week 6: number analyzed (Face sides) | 10 | 10
  Week 6 | -0.7 (7.92) | -0.6 (7.24)
  Week 7: number analyzed (Participants) | 10 | 10
  Week 7: number analyzed (Face sides) | 10 | 10
  Week 7 | 0.8 (6.28) | -1.7 (7.29)

9. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event is any untoward medical occurrence associated with the use of a drug in participants, whether or not considered drug related.
Time Frame: Day 1 until Week 7 (End of Study) and Unscheduled Visit
Population: Safety population included all randomized participants who received test article and applied at least one application.
Measure: Number; unit: Participants
Arm/Group | Overall
Number analyzed (Participants) | 12
Participants
  Any TEAEs | 5
  Any Treatment Related TEAEs | 0
  TEAEs Within the Treatment Area | 0
  Serious TEAEs | 0

10. Primary Outcome: Number of Participants Having Local Skin Reactions With Improved/Same Versus Worsened Severities Compared to Baseline
Description: The local skin reactions (LSRs) included erythema, edema, scaling/dryness, burning/stinging, pruritus, erosion, and pain) were assessed. Erythema, edema, scaling/dryness, and erosion were assessed by the investigator and burning/stinging, pain, and pruritus were assessed by the participant. Assessments was made using a 4-point ordinal scale where 0=absent, 1=mild (slight, barely perceptible), 2=moderate (distinct presence), and 3=severe (marked, intense). Here, lower point represented no reaction and higher points represented severe reactions.The LSRs were assessed both before and 15 minutes following test article application.
Time Frame: Day 1 until Week 7 (End of Study) or Unscheduled Visit
Population: Safety population included all randomized participants who received test article and applied at least one application. Here, overall number of participants analyzed presents only those participants who were analyzed for particular outcome measure, and number analyzed presents the number of participants that were analyzed at specified week.
Measure: Count of Participants; unit: Participants
Arm/Group | FMX101 Oil Vehicle (A) | Hydro-alcohol Vehicle (B)
Number analyzed (Participants) | 11 | 11
Participants
  Erythema, Week 1 (Improved/Same): number analyzed (Participants) | 10 | 10
  Erythema, Week 1 (Improved/Same) | 9 | 9
  Erythema, Week 1 (Worsened): number analyzed (Participants) | 10 | 10
  Erythema, Week 1 (Worsened) | 1 | 1
  Erythema, Week 2 (Improved/Same) | 11 | 11
  Erythema, Week 2 (Worsened) | 0 | 0
  Erythema, Week 4 (Improved/Same): number analyzed (Participants) | 9 | 9
  Erythema, Week 4 (Improved/Same) | 9 | 9
  Erythema, Week 4 (Worsened): number analyzed (Participants) | 9 | 9
  Erythema, Week 4 (Worsened) | 0 | 0
  Erythema, Week 6 (Improved/Same): number analyzed (Participants) | 10 | 10
  Erythema, Week 6 (Improved/Same) | 10 | 10
  Erythema, Week 6 (Worsened): number analyzed (Participants) | 10 | 10
  Erythema, Week 6 (Worsened) | 0 | 0
  Erythema, Week 7 (Improved/Same) | 11 | 11
  Erythema, Week 7 (Worsened) | 0 | 0
  Edema, Week 1 (Improved/Same): number analyzed (Participants) | 10 | 10
  Edema, Week 1 (Improved/Same) | 10 | 10
  Edema, Week 1 (Worsened): number analyzed (Participants) | 10 | 10
  Edema, Week 1 (Worsened) | 0 | 0
  Edema, Week 2 (Improved/Same) | 11 | 11
  Edema, Week 2 (Worsened) | 0 | 0
  Edema, Week 4 (Improved/Same): number analyzed (Participants) | 9 | 9
  Edema, Week 4 (Improved/Same) | 9 | 9
  Edema, Week 4 (Worsened): number analyzed (Participants) | 9 | 9
  Edema, Week 4 (Worsened) | 0 | 0
  Edema, Week 6 (Improved/Same): number analyzed (Participants) | 10 | 10
  Edema, Week 6 (Improved/Same) | 10 | 10
  Edema, Week 6 (Worsened): number analyzed (Participants) | 10 | 10
  Edema, Week 6 (Worsened) | 0 | 0
  Edema, Week 7 (Improved/Same) | 11 | 11
  Edema, Week 7 (Worsened) | 0 | 0
  Scaling/Dryness, Week 1 (Improved/Same): number analyzed (Participants) | 10 | 10
  Scaling/Dryness, Week 1 (Improved/Same) | 10 | 9
  Scaling/Dryness, Week 1 (Worsened): number analyzed (Participants) | 10 | 10
  Scaling/Dryness, Week 1 (Worsened) | 0 | 1
  Scaling/Dryness, Week 2 (Improved/Same) | 9 | 8
  Scaling/Dryness, Week 2 (Worsened) | 2 | 3
  Scaling/Dryness, Week 4 (Improved/Same): number analyzed (Participants) | 9 | 9
  Scaling/Dryness, Week 4 (Improved/Same) | 9 | 9
  Scaling/Dryness, Week 4 (Worsened): number analyzed (Participants) | 9 | 9
  Scaling/Dryness, Week 4 (Worsened) | 0 | 0
  Scaling/Dryness, Week 6 (Improved/Same): number analyzed (Participants) | 10 | 10
  Scaling/Dryness, Week 6 (Improved/Same) | 9 | 8
  Scaling/Dryness, Week 6 (Worsened): number analyzed (Participants) | 10 | 10
  Scaling/Dryness, Week 6 (Worsened) | 1 | 2
  Scaling/Dryness, Week 7 (Improved/Same) | 10 | 11
  Scaling/Dryness, Week 7 (Worsened) | 1 | 0
  Erosion, Week 1 (Improved/Same): number analyzed (Participants) | 10 | 10
  Erosion, Week 1 (Improved/Same) | 10 | 10
  Erosion, Week 1 (Worsened): number analyzed (Participants) | 10 | 10
  Erosion, Week 1 (Worsened) | 0 | 0
  Erosion, Week 2 (Improved/Same) | 11 | 11
  Erosion, Week 2 (Worsened) | 0 | 0
  Erosion, Week 4 (Improved/Same): number analyzed (Participants) | 9 | 9
  Erosion, Week 4 (Improved/Same) | 9 | 9
  Erosion, Week 4 (Worsened): number analyzed (Participants) | 9 | 9
  Erosion, Week 4 (Worsened) | 0 | 0
  Erosion, Week 6 (Improved/Same): number analyzed (Participants) | 10 | 10
  Erosion, Week 6 (Improved/Same) | 10 | 10
  Erosion, Week 6 (Worsened): number analyzed (Participants) | 10 | 10
  Erosion, Week 6 (Worsened) | 0 | 0
  Erosion, Week 7 (Improved/Same) | 11 | 11
  Erosion, Week 7 (Worsened) | 0 | 0
  Burning/Stinging, Week 1 (Improved/Same): number analyzed (Participants) | 10 | 10
  Burning/Stinging, Week 1 (Improved/Same) | 10 | 10
  Burning/Stinging, Week 1 (Worsened): number analyzed (Participants) | 10 | 10
  Burning/Stinging, Week 1 (Worsened) | 0 | 0
  Burning/Stinging, Week 2 (Improved/Same) | 11 | 10
  Burning/Stinging, Week 2 (Worsened) | 0 | 1
  Burning/Stinging, Week 4 (Improved/Same): number analyzed (Participants) | 9 | 9
  Burning/Stinging, Week 4 (Improved/Same) | 9 | 9
  Burning/Stinging, Week 4 (Worsened): number analyzed (Participants) | 9 | 9
  Burning/Stinging, Week 4 (Worsened) | 0 | 0
  Burning/Stinging, Week 6 (Improved/Same): number analyzed (Participants) | 10 | 10
  Burning/Stinging, Week 6 (Improved/Same) | 10 | 10
  Burning/Stinging, Week 6 (Worsened): number analyzed (Participants) | 10 | 10
  Burning/Stinging, Week 6 (Worsened) | 0 | 0
  Burning/Stinging, Week 7 (Improved/Same) | 11 | 11
  Burning/Stinging, Week 7 (Worsened) | 0 | 0
  Pain, Week 1 (Improved/Same): number analyzed (Participants) | 10 | 10
  Pain, Week 1 (Improved/Same) | 10 | 10
  Pain, Week 1 (Worsened): number analyzed (Participants) | 10 | 10
  Pain, Week 1 (Worsened) | 0 | 0
  Pain, Week 2 (Improved/Same) | 11 | 11
  Pain, Week 2 (Worsened) | 0 | 0
  Pain, Week 4 (Improved/Same): number analyzed (Participants) | 9 | 9
  Pain, Week 4 (Improved/Same) | 9 | 9
  Pain, Week 4 (Worsened): number analyzed (Participants) | 9 | 9
  Pain, Week 4 (Worsened) | 0 | 0
  Pain, Week 6 (Improved/Same): number analyzed (Participants) | 10 | 10
  Pain, Week 6 (Improved/Same) | 10 | 10
  Pain, Week 6 (Worsened): number analyzed (Participants) | 10 | 10
  Pain, Week 6 (Worsened) | 0 | 0
  Pain, Week 7 (Improved/Same) | 11 | 11
  Pain, Week 7 (Worsened) | 0 | 0
  Pruritus, Week 1 (Improved/Same): number analyzed (Participants) | 10 | 10
  Pruritus, Week 1 (Improved/Same) | 10 | 10
  Pruritus, Week 1 (Worsened): number analyzed (Participants) | 10 | 10
  Pruritus, Week 1 (Worsened) | 0 | 0
  Pruritus, Week 2 (Improved/Same) | 11 | 11
  Pruritus, Week 2 (Worsened) | 0 | 0
  Pruritus, Week 4 (Improved/Same): number analyzed (Participants) | 9 | 9
  Pruritus, Week 4 (Improved/Same) | 9 | 9
  Pruritus, Week 4 (Worsened): number analyzed (Participants) | 9 | 9
  Pruritus, Week 4 (Worsened) | 0 | 0
  Pruritus, Week 6 (Improved/Same): number analyzed (Participants) | 10 | 10
  Pruritus, Week 6 (Improved/Same) | 10 | 10
  Pruritus, Week 6 (Worsened): number analyzed (Participants) | 10 | 10
  Pruritus, Week 6 (Worsened) | 0 | 0
  Pruritus, Week 7 (Improved/Same) | 11 | 11
  Pruritus, Week 7 (Worsened) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 until Week 7 (End of Study) or Unscheduled Visit
Description: Adverse Events were only monitored/assessed on the whole participant level.
Arm/Group | Overall
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall (N=12)
Gastroenteritis Viral (Gastrointestinal disorders) | 1
Influenza (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT03743038/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/38/NCT03743038/SAP_001.pdf